CLINICAL TRIAL: NCT04781764
Title: The Study of Microglia/Macrophages Involved Dynamic Evolution of Glioma Microenvironment and the Function and Visualization of Targeted Molecules of Glioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yu Yao, MD, Professor, Huashan Hospital
Other Study IDs: KY2020-009
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- glioma patients: glioma patients with routine surgery
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — surgery

SUMMARY:
establishment of glioma microenvironment cell dynamic evolution database reveal the mechanism of GIM promoting malignant transformation of glioma cells reveal the dynamic regulation process of immune cells in the process of glioma evolution

DETAILED DESCRIPTION:
To collect tissue samples from different stages of glioma evolution and establish a high-quality high-throughput sequencing database of immune microenvironment cells, so as to lay a data foundation for later mining the dialogue mechanism and key targets between immune cells and tumor cells in glioma microenvironment.

Based on the analysis results of the above database, the key role of key target molecules in the dialogue between GIM and glioma cells and the regulation ability of immune cells in the immune microenvironment were confirmed through cell and mouse animal experiments, which laid the foundation for later targeted drug research and development.

Combined with fluorescence imaging technology, through in vivo imaging of mice, it can provide more intuitive and effective visual verification for the dynamic infiltration process of GIM and other immune microenvironment cells in the process of glioma evolution, and provide a new theoretical basis for the visualization research of dynamic regulation of glioma immune microenvironment cells.

ELIGIBILITY:
Inclusion Criteria:

* The patients with glioma in the Department of Neurosurgery of Huashan Hospital Affiliated to Fudan University who meet the following three conditions can be enrolled

  1. They were 18-80 years old, male and female;
  2. The pathological results of frozen section during operation were gliomas (20 cases of who grade II, II and IV, respectively);
  3. Tissue (6 mm * 6 mm) can be used for cell sorting on the basis of not affecting clinical routine diagnosis;
  4. Sign informed consent.

Exclusion Criteria:

* Patients who meet any of the following criteria will not be included in this study:

  1. Participants in other clinical trials;
  2. Pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing glioma surgery at Huashan Hospital
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Multi-omics characteristics of glioma patients | 24 month
  we aim to describe patient's features about transcriptomics 、Immunomics、Radiomics ，etc.
expression level of protein，drived from paraffin-embedded specimens， retrospectively collected. | 24 month
  different expression level of proteins in Gliomas with different grades and molecular subgroups (500 cases)

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital，Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostrom QT, Gittleman H, Farah P, Ondracek A, Chen Y, Wolinsky Y, Stroup NE, Kruchko C, Barnholtz-Sloan JS. CBTRUS statistical report: Primary brain and central nervous system tumors diagnosed in the United States in 2006-2010. Neuro Oncol. 2013 Nov;15 Suppl 2(Suppl 2):ii1-56. doi: 10.1093/neuonc/not151. No abstract available. PMID 24137015
- [Background] Wicki A, Mandala M, Massi D, Taverna D, Tang H, Hemmings BA, Xue G. Acquired Resistance to Clinical Cancer Therapy: A Twist in Physiological Signaling. Physiol Rev. 2016 Jul;96(3):805-29. doi: 10.1152/physrev.00024.2015. PMID 27142452
- [Background] Ribas A, Wolchok JD. Cancer immunotherapy using checkpoint blockade. Science. 2018 Mar 23;359(6382):1350-1355. doi: 10.1126/science.aar4060. Epub 2018 Mar 22. PMID 29567705
- [Background] Chen DS, Mellman I. Oncology meets immunology: the cancer-immunity cycle. Immunity. 2013 Jul 25;39(1):1-10. doi: 10.1016/j.immuni.2013.07.012. PMID 23890059
- [Background] Gotwals P, Cameron S, Cipolletta D, Cremasco V, Crystal A, Hewes B, Mueller B, Quaratino S, Sabatos-Peyton C, Petruzzelli L, Engelman JA, Dranoff G. Prospects for combining targeted and conventional cancer therapy with immunotherapy. Nat Rev Cancer. 2017 May;17(5):286-301. doi: 10.1038/nrc.2017.17. Epub 2017 Mar 24. PMID 28338065
- [Background] Kim PS, Armstrong TD, Song H, Wolpoe ME, Weiss V, Manning EA, Huang LQ, Murata S, Sgouros G, Emens LA, Reilly RT, Jaffee EM. Antibody association with HER-2/neu-targeted vaccine enhances CD8 T cell responses in mice through Fc-mediated activation of DCs. J Clin Invest. 2008 May;118(5):1700-11. doi: 10.1172/JCI34333. PMID 18398507
- [Background] Peng W, Chen JQ, Liu C, Malu S, Creasy C, Tetzlaff MT, Xu C, McKenzie JA, Zhang C, Liang X, Williams LJ, Deng W, Chen G, Mbofung R, Lazar AJ, Torres-Cabala CA, Cooper ZA, Chen PL, Tieu TN, Spranger S, Yu X, Bernatchez C, Forget MA, Haymaker C, Amaria R, McQuade JL, Glitza IC, Cascone T, Li HS, Kwong LN, Heffernan TP, Hu J, Bassett RL Jr, Bosenberg MW, Woodman SE, Overwijk WW, Lizee G, Roszik J, Gajewski TF, Wargo JA, Gershenwald JE, Radvanyi L, Davies MA, Hwu P. Loss of PTEN Promotes Resistance to T Cell-Mediated Immunotherapy. Cancer Discov. 2016 Feb;6(2):202-16. doi: 10.1158/2159-8290.CD-15-0283. Epub 2015 Dec 8. PMID 26645196
- [Background] Syed Khaja AS, Toor SM, El Salhat H, Faour I, Ul Haq N, Ali BR, Elkord E. Preferential accumulation of regulatory T cells with highly immunosuppressive characteristics in breast tumor microenvironment. Oncotarget. 2017 May 16;8(20):33159-33171. doi: 10.18632/oncotarget.16565. PMID 28388539
- [Background] Watters JJ, Schartner JM, Badie B. Microglia function in brain tumors. J Neurosci Res. 2005 Aug 1;81(3):447-55. doi: 10.1002/jnr.20485. PMID 15959903